CLINICAL TRIAL: NCT00570544
Title: Effectiveness of Tiotropium to Maintain Inspiratory Capacity Against Metronome Paced Hyperventilation Induced Dynamic Hyperinflation in COPD Patients With Lung CT Scored Emphysema
Brief Title: Tiotropium Induced Bronchodilation in Lung CT Scored Emphysema
Status: Completed | Type: Observational
Sponsor: Gelb, Arthur F., M.D. (Individual)
Collaborators: Boehringer Ingelheim (Industry); Pfizer (Industry)
Responsible Party: Arthur F Gelb MD, Arthur F Gelb Medical Corporation
Other Study IDs: 1000; Boehringer-Ingelheim Pharm.; Pfizer
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2008-08-14 (Estimated); Status verified 2007-12

CONDITIONS: COPD; Emphysema
Keywords: copd; emphysema; tiotropium; lung function; dynamic hyperinflation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: patients with moderate to severe copd with varying extent of emphysema
  Interventions: Drug: tiotropium

INTERVENTIONS:
Drug: tiotropium — 18ug capsule daily for 30 days
  Other Names: Spiriva

SUMMARY:
To evaluate if tiotropium (Spiriva)induced bronchodilation of inspiratory capacity in patients with moderate to severe copd subjected to metronome paced hyperventilation induced dynamic hyperinflation is dependent upon the extent of underlying emphysema as determined by high resolution-thin section CT lung.

DETAILED DESCRIPTION:
We will analyze post hoc, data that was previously published: Gelb AF et al.Chest 2006;131:690-695. We have shown that tiotropium increases resting inspiratory capacity thereby providing lung volume protection against metronome paced hyperventilation induced dynamic hyperinflation. End point will be to correlate increase in tiotropium induced FEV 1(L) and inspiratory capacity with extent of underlying emphysema as scored by lung CT ( Gelb AF et al:Chest 1996; 109: 353-359)in 29 patients with COPD. We will also correlate the decrease in inspiratory capacity following metronome paced hyperventilation induced dynamic hyperinflation with extent of lung CT scored emphysema.

ELIGIBILITY:
Inclusion Criteria

* moderate to severe copd

Exclusion Criteria

* unable to tolerate tiotropium
* unable to perform metronome paced hyperventilation induced dynamic hyperinflation

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with moderate to severe copd from tertiary care pulmonary clinic
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2004-08; Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Correlate tiotropium induced increase in inspiratory capacity (IC)and FEV 1 with extent of emphysema as scored by lung CT. | After 30 days and 1.5hr of tiotropium

SECONDARY OUTCOMES:
Correlate decrease in IC and FEV 1 following dynamic hyperinflation with underlying emphysema. | After 30 days and 1.5hr of tiotropium

CONTACTS AND LOCATIONS:
Overall Officials: Arthur F Gelb, MD, Principal Investigator — Arthur F Gelb Medical Corporation
Locations (1):
- Arthur F Gelb Medical Corporation, Lakewood, California, United States

REFERENCES:
- [Background] Gelb AF, Taylor CF, McClean PA, Shinar CM, Rodrigues MT, Gutierrez CA, Chapman KR, Zamel N. Tiotropium and simplified detection of dynamic hyperinflation. Chest. 2007 Mar;131(3):690-695. doi: 10.1378/chest.06-1662. PMID 17356081
- [Background] Gelb AF, Hogg JC, Muller NL, Schein MJ, Kuei J, Tashkin DP, Epstein JD, Kollin J, Green RH, Zamel N, Elliott WM, Hadjiaghai L. Contribution of emphysema and small airways in COPD. Chest. 1996 Feb;109(2):353-9. doi: 10.1378/chest.109.2.353. PMID 8620705